CLINICAL TRIAL: NCT07026058
Title: Effects Of Sound Sine Wave And Standard Physiotherapy On Pain, Mobility, Function And Pelvic Alignment In Mechanical Low Back Pain
Brief Title: Sound Sine Wave And Standard Physiotherapy In Mechanical Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Aleena- REC/RCR&AHS 24/0135
Record Dates: First submitted 2025-06-11; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Low Back Pain
Keywords: Low Back Pian; Physical Therapy; Disability; Pelvic Alignment; Range of Motion; Pain
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Other: Sound Wave Treatment
- Group B (Active Comparator)
  Interventions: Other: Standard physiotherapy

INTERVENTIONS:
Other: Sound Wave Treatment — Sound wave treatment with 6 sessions initially, 3 times a week, followed by the next 6 sessions with a frequency of 2 times a week. Patient's position was analysed through digital X-ray of cervical spine, 80 pulses are typically administered in a session. These pulses are applied generally, targeting the 1st cervical vertebra of the spine. This method aims to achieve spinal alignment through the vibrations generated by the treatment. Before and after the treatment, a patient assessment is conducted to observe visible improvements. A mixed waveform of 8Hz-202 Hz resonated throughout the spine, with intensities ranging from 0.3 to 1. In order to affect the lumbar region, where they are also applied, sound waves are employed to activate C1.
  After First 3 sessions vibrations on pain focal points also given to the patient the 40 pulses are typically administrated at pain point.
  Arms: Group A
Other: Standard physiotherapy — Flexibility Training: Stretching exercises are crucial to improve the flexibility of the spine and surrounding muscles. This includes stretches for the hamstrings, hip flexors, and lower back Strengthening Exercises: Focus on strengthening the core muscles, including the abdominal and back muscles. Common exercises include pelvic tilts, bridging, and lumbar stabilization exercises Postural Training: Education and exercises to correct posture are vital. Proper posture reduces strain on the spine and helps prevent further injury.(31). Techniques such as ergonomic adjustments at work and home, along with exercises like seated squats and calf stretches Manual Therapy: Techniques such as myofascial release (32) and spinal mobilization. Spinal mobilization as one of the most preferable approaches for the management of LBP
  Arms: Group B

SUMMARY:
The study design will be a randomized clinical trial (RCT). Sampling technique will be nonprobability convenience sampling. Data will be collected from KKT orthopedic spine center Lahore. Participants will be divided into 2 groups. Group A will receive Sound wave treatment protocol and standard physiotherapy treatment protocol , Group B will receive only Standard Physiotherapy treatment .Both groups will receive TENS and hot pack for 10 minutes. The inclusion and exclusion criteria will be Both gender , aged 18-45 years , Minimum 03 months chronicity of lower back pain , Clinically diagnosed with the help of tests SLR test to rule out nerve root compression or disc herniation, FABER test to rule out SI joint dysfunction ,Scobber Test to assess lumbar flexibility and mobility, Lumber quadrant test to identify pain from facet joints, Lumber extension test and Pain localized to the lumbar region, potentially radiating to the buttocks or thighs but not below the knee. The Exclusion Criteria will be Chronic systemic soft tissue and bony diseases , History of spinal trauma or fractures , Severe spinal stenosis or spondylolisthesis and Pain radiating to one or both legs, consistent with lumbar radiculopathy. The outcome measure tools will be NPRS, inclinometer, x-rays and Oswestry Disability Index (ODI) . Data will be analyzed using SPSS . Ethical Committee of Riphah International University, and informed consent will be secured from all participants.

DETAILED DESCRIPTION:
Low back pain (LBP) is considered one of the most common musculoskeletal disorders that affect people of all ages around the world. In addition, LBP is becoming a burden in many developing and low-income countries due to high healthcare costs for its treatment and management. Low back pain (LBP) is defined as a pain or discomfort located below the margin of the 12th rib and above the inferior gluteal fold, with or without leg pain. Low back pain covers a spectrum of different types of pain (eg, nociceptive, neuropathic and nociplastic, or non-specific) that frequently overlap. The elements comprising the lumbar spine (eg, soft tissue, vertebrae, zygapophyseal and sacroiliac joints, intervertebral discs, and neurovascular structures) are prone to different stressors, and each of these, alone or in combination, can contribute to low back pain. Low back pain (LBP) is a highly prevalent and complex condition. It is associated with significant socio-economic costs. Currently, it is the leading cause of disability worldwide. Most episodes of LBP resolve within 6 weeks but 10-15% become chronic. People more often leave their job because of low back pain than diabetes, hypertension, neoplasm, asthma, heart and respiratory disease combined. More than 85% of LBP cases are categorized as nonspecific LBP (NSLBP) with no identifiable cause or pathology. Postural control, which is essential for executing functional activities, is diminished in patients with NSLBP . Chronic low back pain (CLBP) is a complex and multifactorial musculoskeletal disorder (MSKD) that has become the leading cause of disability worldwide. According to the Global Burden of Disease 2017, the years lived with disability (YLD) due to LBP increased by 52.7%, from 42.5 million in 1990 to 64.9 million in 2017. In 2019, the global LBP prevalent cases were 568.4 million, with an age standardized point-prevalence of 6972.5 per 100,000 population and 223.5 million incidence cases with an age-standardized annual incidence of 2748.9, globally. Low back pain (LBP) is the leading cause of years lived in disability in high-income and middle-income countries. Moreover, a similar increase has also been seen in low-income countries. Musculoskeletal disorders contribute about 3.4% and 1.7% of the total global burden of disease in highincome-countries and low-and-middle-income-countries, respectively.

The study aims to investigate the combined effects of sound sine wave therapy and standard physiotherapy on mechanical low back pain. This approach is rooted in the idea of enhancing conventional physiotherapy outcomes by exploring the potential benefits of sound therapy, which may include pain relief, improved mobility, restored function, and corrected pelvic alignment. By integrating these modalities, the study seeks to contribute empirical evidence to support their complementary roles in managing chronic low back pain and optimizing musculoskeletal rehabilitation strategies

ELIGIBILITY:
Inclusion Criteria:

* Both gender Aged 18-45 years
* Minimum 03 months chronicity of lower back pain
* Clinically diagnosed with the help of tests
* SLR test to rule out nerve root compression or disc herniation
* FABER test to rule out SI joint dysfunction
* Scobber Test to assess lumbar flexibility and mobility
* Lumber quadrant test to identify pain from facet joints
* Lumber extension test
* Pain localized to the lumbar region, potentially radiating to the buttocks or thighs but not below the knee

Exclusion Criteria:

* Chronic systemic soft tissue and bony diseases
* History of spinal trauma or fractures
* Severe spinal stenosis or spondylolisthesis
* Pain radiating to one or both legs, consistent with lumbar radiculopathy
* Participants with a known history of cervical myelopathy, characterized by symptoms of spinal cord compression in the cervical spine (e.g., neck pain with neurological deficits such as weakness, numbness, or abnormal reflexes)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-28 (Estimated)

PRIMARY OUTCOMES:
NPRS | Baseline, 4th Week
Oswetry Disability Index | Baseline, 4th Week
Lubmbar Range of Motion | Baseline, 4th Week

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil ur Rehman, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Knezevic NN, Candido KD, Vlaeyen JWS, Van Zundert J, Cohen SP. Low back pain. Lancet. 2021 Jul 3;398(10294):78-92. doi: 10.1016/S0140-6736(21)00733-9. Epub 2021 Jun 8. PMID 34115979
- [Background] Hawamdeh M, Altaim TA, Shallan A, Gaowgzeh RA, Obaidat SM, Alfawaz S, Al-Nassan SM, Neamatallah Z, Eilayyan O, Alabasi UM, Albadi M. Low Back Pain Prevalence among Distance Learning Students. Int J Environ Res Public Health. 2022 Dec 26;20(1):342. doi: 10.3390/ijerph20010342. PMID 36612660